CLINICAL TRIAL: NCT00397449
Title: Assessment of the Safety and Immunogenicity of the Recombinant Lactococcus Lactis Hybrid GMZ2 [GLURP+MSP3] a Malaria Vaccine in Healthy Adult Volunteers. A Phase I, Double-Blind, Randomised, Dose-Selection, Unicentre Trial
Brief Title: GMZ2-Aluminum Hydroxide Phase I, Tübingen
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Vaccine Initiative (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EudraCT: 2005-004568-22
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Malaria
Keywords: Malaria, malaria vaccine, randomised, safety, immunogenicity
MeSH Terms: conditions — Malaria | interventions — Malaria Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, 2, 3 (Experimental)
  Interventions: Biological: GMZ2 (GLURP + MSP3 Hybrid) (malaria vaccine)

INTERVENTIONS:
Biological: GMZ2 (GLURP + MSP3 Hybrid) (malaria vaccine)

SUMMARY:
This is a randomized, open, dose-selection Phase 1 study. The study aims to evaluate the safety and immunogenicity of 3 doses (10,30 & 100 micrograms) of the GMZ2 hybrid (GLURP and MSP3) blood stage vaccine in healthy non-immune European adults. The vaccines will be administered with aluminum hydroxide as adjuvant. The safety and the tolerability of the vaccine will be assessed on the rate of solicited and unsolicited events/reactions related to the vaccine. The safety profile will include local and systemic reactions/events as well as the biological safety, based on a clinically significant change of the baseline value of the main biological criteria. The immunogenicity of the different formulation of the vaccine will be assessed on the level and the quality of circulating antibodies as well as the stimulation of the T-cell immune response.

DETAILED DESCRIPTION:
The trial is a randomised, open, dose-selection, single centre trial. One adjuvant will be assessed, aluminum hydroxide (alum). Three different dosages - 10µg, 30µg, and 100µg - of GMZ2 will be evaluated with the aluminum hydroxide adjuvant. A total of 30 volunteers will be enrolled and randomized into three groups of 10. As this is a dose escalation study, volunteers in Group 1 will receive the initial dose of 10µg on the first vaccination day. After a satisfactory safety profile at this dose (see sections 6.2.2 and 6.2.3), we will proceed to vaccinate volunteers in Group 2 with the higher dose of 30µg after a 2-week interval. The same procedure will also be followed for volunteers in Group 3, who will be administered their initial dose of 100µg GMZ2 if the review of the safety profile of Group 2 is satisfactory. The aim will be to recruit all volunteers before the intended start of the study. The randomization procedure will be performed in the following way: when participants are found to be eligible and have signed their informed consent they will be numbered sequentially (in order of enrollment). The numbers will be randomly assigned to 3 groups of 10 numbers through a specific randomization computer program. These groups will be the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 45 years healthy volunteers (males or females)
* General good health based on history and clinical examination
* All volunteers have to sign the informed consent form
* Negative pregnancy test
* Use of adequate contraception for females up to three months after the third injection (D140)
* Intention to not travel abroad and reachable by phone during the whole study period (15 months).

Exclusion Criteria:

* History of malaria or residence in malaria endemic areas for the past six months.
* Positive serology for malaria antigen GLURP and/or MSP3.
* Previously participated in a malaria vaccine studies.
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Any laboratory abnormalities on screened blood samples beyond the normal range, as defined at Tübingen. Positive HIV, HBV or HCV tests
* Volunteers should not be enrolled in any other clinical trial during the whole trial period
* Volunteers should not receive chronic medication, especially immunosuppressive agents (steroids, immuno-modulating or immunosuppressive drugs) during the three months preceding the screening visit or during the study period
* Pregnant or lactating women
* Volunteers unable to give written informed consent
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrollment in the study
* Volunteers should not perform exercise four hours before blood draw and should not donate blood for non study-related purposes during the entire duration of the study
* Known hypersensitivity to any of the vaccine components (adjuvant or peptide)
* Volunteers are not allowed to receive any vaccination or gammaglobulin during a period three months prior to the first immunization and up to six months after the 3rd immunization. If a vaccination is necessary during this period, the volunteer will be withdrawn from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Safety | one year
Immunogenicity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Knobloch, MD, Principal Investigator — Insitut of Tropical Medicine, University of Tubingen; Peter Kremsner, MD, PhD, Study Director — Insitut of Tropical Medicine, University of Tubingen
Locations (1):
- Institut for Tropical Medicine, University of Tubingen, Tübingen, Germany

REFERENCES:
- See also: website of the European Malaria Vaccine Initiative — http://www.emvi.org